CLINICAL TRIAL: NCT07178119
Title: A Prospective Clinical Evaluation of the Bridging Technique Using AILEENE Vol. 2 Dermal Filler for the Treatment of Nasolabial Folds
Brief Title: Bridging Technique Validation for Nasolabial Folds JN-BRIDGE-1
Acronym: BRIDGING
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Joseph M Novoa Libermann (Other)
Collaborators: Cg Bio Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Dr. Joseph M Novoa Libermann, Principal Investigator, JNL Aesthetics Limited
Organization: JNL Aesthetics Limited (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JNL-BridgingNL-2025; JNL-BridgingNL-2025 (Registry Identifier: IRAS)
Record Dates: First submitted 2025-08-31; First posted 2025-09-17 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Nasolabial Fold Correction; Facial Aging; Skin Rejuvenation; Wrinkles Such as Nasolabial Folds
Keywords: Hyaluronic Acid Filler; Dermal Filler; AILEENE Vol. 2; Bridging Technique; Minimally Invasive Aesthetics; Non-Surgical Facial Rejuvenation; Wrinkle Correction; Global Aesthetic Improvement Scale (GAIS); Nasolabial Fold Severity Scale (NLFSS)

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-arm clinical evaluation study of the Bridging Technique using AILEENE Vol. 2 hyaluronic acid (HA) dermal filler for the correction of nasolabial folds (NLF). All enrolled participants will receive the same intervention.
Masking Description: This is a prospective, single-arm study and is therefore registered as Open Label. Participant, care provider, and investigator masking is not possible. However, outcome assessment is blinded. Standardized photographs obtained at Baseline (Day 0), Week 4, Month 3, and Month 6 will be evaluated by two independent observers who are not involved in treatment or follow-up. Observers are blinded to participant identity and to the chronological order of images; discrepancies are resolved by consensus. A virtual safety check is performed at Week 2; no formal outcome scoring occurs at this time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bridging Technique with AILEENE Vol. 2 (Experimental): Although AILEENE Vol. 2 is a hyaluronic acid (HA) dermal filler that is Conformité Européenne (CE)-marked and registered with the Medicines and Healthcare products Regulatory Agency (MHRA) for use in routine aesthetic practice, the Bridging Technique for the correction of nasolabial folds (NLF) has not yet been formally evaluated in a structured clinical study. For this reason, the intervention is designated as Experimental in this trial.
  Interventions: Procedure: (Bridging) Horizontal Cannula Technique for Treatment of Nasolabial Folds using AILEENE Vol. 2

INTERVENTIONS:
Procedure: (Bridging) Horizontal Cannula Technique for Treatment of Nasolabial Folds using AILEENE Vol. 2 — Participants will receive treatment to both NLF using the Bridging Technique. This involves injecting an HA dermal filler (AILEENE Vol. 2) in thin horizontal threads (less than 0.05 milliliters [ml] per retrograde placement) under the fold using a blunt cannula. The maximum total dose per participant is 1.0 ml across both folds. Each participant will receive one treatment at baseline (Day 0). An optional single top-up may be given at Week 2 (virtual or in-clinic) or Week 4 if clinically indicated, using only the remaining balance of the 1.0 ml total. Any top-up will be performed with a new, sterile syringe, not with filler left over from the initial treatment. This is a single-treatment course with follow-up for 6 months. Standardized photographs will be taken at Baseline, Week 4, Month 3, and Month 6 for blinded assessment.
  Other Names: Bridging Technique for Nasolabial Folds; Horizontal Cannula Injection for Nasolabial Folds; Cannula Technique for Nasolabial Folds; AILEENE Vol. 2; Hyaluronic Acid Dermal Filler; HA Filler

SUMMARY:
The goal of this clinical study is to learn whether the Bridging Technique can safely and effectively treat nasolabial folds (NLF, also known as smile lines) in adults. The main questions are:

Does the Bridging Technique, which places very small amounts of filler in thin horizontal threads (less than 0.05 milliliters [ml] per retrograde placement), improve the appearance of nasolabial folds?

Is the treatment safe, and are participants satisfied with the results?

The Bridging Technique is a new method of filler injection where very small amounts of hyaluronic acid (HA) filler are placed in thin horizontal lines under the fold using a blunt cannula. These small "bridges" of filler act like internal support, helping to lift and soften the fold without overfilling or distorting the natural shape of the face.

Participants will:

Receive an HA dermal filler (AILEENE Vol. 2) injected with the Bridging Technique to both nasolabial folds.

Attend follow-up visits at Week 2 (virtual safety check), Week 4, Month 3, and Month 6.

Have photographs taken at baseline, Week 4, Month 3, and Month 6, which will be reviewed by independent observers who are blinded to the visit sequence.

Complete short questionnaires about their satisfaction and experience.

The study includes 60 adults aged 30 to 65 years. Each participant may receive up to 1.0 ml of filler in total across both folds. An optional top-up treatment may be offered at Week 2 or Week 4 if clinically indicated, using only the remaining balance of the total 1.0 ml allowance. Any top-up will be performed with a new, sterile syringe, not with filler physically left over from the first visit. There is no cost to participants, and participation is voluntary.

DETAILED DESCRIPTION:
Nasolabial folds (NLF) are a visible sign of facial aging and one of the most frequent concerns expressed by patients seeking non-surgical facial rejuvenation. These folds develop due to natural changes in skin elasticity, soft tissue support, and fat distribution. Many patients now request outcomes that are natural in appearance, rather than overly augmented, and wish to achieve this with the least amount of product and downtime.

The Bridging Technique was developed by Dr. Joseph Novoa Libermann in response to this clinical demand. The technique involves the placement of small threads of HA filler across the nasolabial folds using a cannula introduced through a single entry point. This approach is intended to minimize trauma, reduce the risk of vascular compromise (VC), and provide visible improvement with reduced filler volume compared to more traditional methods.

Although the method has been applied in aesthetic practice for over three years with positive results, it has not yet been validated in a structured clinical study. This trial is therefore designed to generate systematic evidence on safety and effectiveness. The focus is on confirming whether the Bridging Technique can consistently achieve natural-looking improvement in nasolabial fold severity while maintaining a favorable safety profile.

The study will also explore the broader impact on patient satisfaction and perceived improvement by combining independent photographic assessment with patient-reported outcome measures (PROMs). By formally documenting outcomes under ethical review and structured follow-up, the study aims to provide clinicians with robust evidence supporting a safer and more conservative approach to nasolabial fold treatment.

The results are intended to support wider adoption of the technique in aesthetic practice, with potential benefits for patient safety, cost-effectiveness, and treatment satisfaction.

ELIGIBILITY:
Inclusion Criteria

Adults aged 30 to 65 years, inclusive, at the time of screening.

Male or female, able and willing to comply with study procedures.

Presence of visible bilateral nasolabial folds (NLF), each with a score of 2 or higher on the Nasolabial Fold Severity Scale (NLFSS), as assessed by the Principal Investigator.

Willing to undergo facial dermal filler treatment using the Bridging Technique with AILEENE Vol. 2.

In generally good health, without uncontrolled chronic illness or active skin disease that could interfere with treatment or healing.

Able to provide written informed consent and understand the nature and purpose of the study.

Willing to refrain from undergoing any other facial cosmetic procedures (e.g., dermal fillers, botulinum toxin, laser, surgery, or radiofrequency) during the six-month study period.

Agree to photographic documentation of the treatment area and follow-up assessments, and willing to allow use of anonymized photographs for blinded evaluation and publication.

For women of childbearing potential: negative urine pregnancy test at baseline.

Female participants of childbearing potential will undergo a urine pregnancy test on the day of treatment as a safety precaution, since there is insufficient evidence on filler safety during pregnancy.

Exclusion Criteria Presence of NLF graded less than 2 on the NLFSS on either side of the face.

Known allergy or hypersensitivity to hyaluronic acid (HA), lidocaine, or any component of AILEENE Vol. 2.

History of severe allergic reactions, anaphylaxis, or allergy to local anesthetics.

Prior use of dermal fillers, permanent implants, or other cosmetic procedures in the NLF area or lower face within the past 12 months.

Use of botulinum toxin, chemical peels, laser, radiofrequency, or cryotherapy in the mid- or lower face within the last six months.

Active skin infection, inflammation, herpes simplex (cold sore), acne, or other dermatologic condition in the treatment area.

Use of topical medications such as retinoids or corticosteroids on the face within 30 days prior to treatment.

Current or recent use (within 14 days) of anticoagulant, antiplatelet, or non-steroidal anti-inflammatory drugs (NSAIDs) that may increase the risk of bruising or bleeding.

History of bleeding disorders.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-22 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change in Nasolabial Fold Severity using the Nasolabial Fold Severity Scale (NLFSS) | Baseline (Day 0), Week 4, Month 3, and Month 6
  The Nasolabial Fold Severity Scale (NLFSS) is a 5-grade photographic severity scale used to rate the depth and appearance of nasolabial folds. It is based on a modified version of the Wrinkle Severity Rating Scale (WSRS), adapted specifically for nasolabial fold evaluation.
  Scale:
  Grade 0 - Absent: No visible fold Grade 1 - Mild: Shallow fold, barely visible indentation Grade 2 - Moderate: Clear fold, moderate indentation Grade 3 - Severe: Deep and prominent fold Grade 4 - Very Severe: Very deep, highly visible fold with sharp demarcation
  Two independent blinded observers will compare baseline and follow-up photographs of each participant against the NLFSS reference images and assign scores. Any discrepancies will be resolved by consensus. Improvement is defined as a decrease in score from baseline.Statistical analysis will use a paired t-test

SECONDARY OUTCOMES:
Change in Aesthetic Appearance using the Global Aesthetic Improvement Scale (GAIS) | Week 4, Month 3, and Month 6
  The Global Aesthetic Improvement Scale (GAIS) is a five-point scale that measures overall aesthetic improvement compared with baseline:
  1. = Very much improved
  2. = Much improved
  3. = Improved
  4. = No change
  5. = Worse
  Two independent blinded observers will assess standardized photographs using the GAIS. Participants will also complete a self-assessment GAIS questionnaire at each follow-up visit.

OTHER OUTCOMES:
Patient Satisfaction and Treatment Experience Using a Five-Item Patient-Reported Outcome Measure (PROM) | Week 4, Month 3, and Month 6
  A five-item questionnaire will be administered using a five-point Likert scale to assess:
  1. -Satisfaction with appearance
  2. -Comfort during treatment
  3. -Perceived improvement
  4. -Willingness to repeat the procedure
  5. -Overall satisfaction
Proportion of Participants Requesting Top-Up Treatment at Week 4 | Week 4
  The proportion of participants who request or receive an optional top-up filler at the Week 4 visit will be documented in the Case Report Forms(CRFs).

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M Novoa Libermann, MBBS, Principal Investigator — JNL Aesthetics Limited
Locations (1):
- JNL Aesthetics Limited, Warrington, Cheshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. This is a single-site aesthetic medicine study with a small sample size (n=60). To protect participant confidentiality, only anonymised summary results will be made publicly available on ClinicalTrials.gov. Study findings will also be submitted for publication in a peer-reviewed scientific journal.

REFERENCES:
- See also: PDF brochure detailing physical and structural properties of AILEENE Vol. 2, including its multi-layered phasic structure and rheological metrics. — https://easyfairsassets.com/sites/188/2023/06/AiLEENE_Hybrid-HA-dermal-filler.pdf
- See also: CG Bio research page. CG Bio is the manufacturer of AILEENE Vol. 2 dermal filler and publishes educational scientific materials, although it is not the study sponsor. — https://www.cgbio.co.kr/en/paper/all
- Available data/document: Study Protocol: JNL-BridgingNL-2025 — https://ascenciaa.com/docs/study-protocol-version-1-0-jnl-bridgingnl-2025/ — The study protocol (Version 1.0, 27 August 2025, REC approved) is publicly available on the sponsor's website, Ascencia Aesthetics Academy. It can be accessed directly via the link above or by navigating to the "About" page under the "Vision" section of the website.

DOCUMENTS (2):
  • Study Protocol (2025-08-01): https://cdn.clinicaltrials.gov/large-docs/19/NCT07178119/Prot_000.pdf
  • Informed Consent Form (2025-08-27): https://cdn.clinicaltrials.gov/large-docs/19/NCT07178119/ICF_001.pdf